CLINICAL TRIAL: NCT06684574
Title: Effects of Covid-19 and Nordic Walking on Older People with Knee Osteoarthritis
Brief Title: Nordic Walking on Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Consorci Hospitalari de Vic (Other)
Responsible Party: Principal Investigator, Dr. Pere Roura-Poch, Philosophy doctor, Consorci Hospitalari de Vic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P153
Record Dates: First submitted 2024-11-08; First posted 2024-11-12 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Osteoarthritis of Knee
Keywords: Knee osteoarthritis; Quality of life; Covid-19; Exercise therapy; Nordic walking
MeSH Terms: conditions — Osteoarthritis, Knee; COVID-19

STUDY DESIGN:
Intervention Model Description: Intervention is a program of nordic walking and strengtheining exercises
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nordic walking program (Active Comparator): Patients randomly allocated this arm participated in a nordic walking program to improve their pain symptoms and quality of life
  Interventions: Other: Nordic walking program
- Control group (Placebo Comparator): Patients randomly assigned to this group received only one educational session to advice the convenience of exercising on their own initiative.
  Interventions: Other: Educational advise

INTERVENTIONS:
Other: Nordic walking program — The intervention is a defined program of Nordic walking and strengthening exercises for 10 weeks in a regimen of two days per week (two 75-minute sessions per week). In these sessions, they did Nordic walking three 5-minute breaks, where strength and proprioception exercises of the lower extremities were performed.
  Arms: Nordic walking program
Other: Educational advise — Patients in the control arm participated in a single session to advise them on the need for self-exercise.
  Arms: Control group

SUMMARY:
The goal of this randomized clinical trial is to improve osteoarthritis symptoms and quality of life in older people with knee osteoarthritis from a primary care center. The main question it aims to answer is:

* To participate in a Nordic walking reduces pain measured on WOMAC pain dimension?
* To participate in a Nordic walking improves mobility measured on WOMAC physical activitiy dimension? Researchers will compare pain and physical activity outcomes between intervention and control arm (randomly allocated).

DETAILED DESCRIPTION:
Osteoarthritis is one of the clinical circumstances that produces the most disability in terms of disability-adjusted life years (DALYs), its main localization is in the knees and hips, the most disabling joints. Ten percent of the adult Spanish population has knee osteoarthritis , which is accompanied by symptoms of pain, mechanical alterations, stiffness, and decreased functionality, constituting one of the most common causes of disability in older people.. Decreased muscle mass and strength of knee extensor-flexor muscles are associated with symptomatic progression of oseoarthritis and lower general health status.

ELIGIBILITY:
Inclusion Criteria:

* Aged of 60 years or older
* Knee osteoarthritis
* Body mass index less than 35 kg/m2

Exclusion Criteria:

* People who had a knee prostheses
* To have any contraindication for physical activity
* To have an acute exacerbation of any chronic condition at enrollment

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Western Ontario and McMaster Universities Osteoarthritis Index | From enrollment to the end of treatment at 10 weeks
  The Western Ontario and McMaster Universities Arthritis Index (WOMAC) is widely used in the evaluation of Hip and Knee Osteoarthritis. It is a self-administered questionnaire consisting of 24 items divided into 3 subscales: pain (5 items), stiffness (2 items) and physical function. WOMAC is available and validated in Spanish language. Overall, the sum of the three dimensions can have a minimum of zero points and a maximum of 96 points where 0 represents the best health status and 96 the worst possible status. The higher the score, the poorer the function.

SECONDARY OUTCOMES:
36-Item Short Form Survey Instrument (SF-36) | From enrollment to the end of treatment at 10 weeks
  The 36-Item Short Form Survey (SF-36) is an outcome measure instrument that is often used, well-researched, self-reported measure of physical and mental health scores. The SF-36 has eight scaled scores; the scores are weighted sums of the questions in each section. Scores range from 0 - 100 where lower scores identifies more disability and higher scores identifies less disability. The sections are vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, emotional role functioning, social role functioning and mental health.

OTHER OUTCOMES:
Time up and go | From enrollment to the end of treatment at 10 weeks
  The test begins with the subject sitting correctly in a chair with arms, the subject's back should resting on the back of the chair. The chair should be stableand positioned such that it will not move when the subject moves from sitting to standing. On the word "go" the subject sou will stand up, walk to the line on the floor (3 meters from the chair), turn around and walk back to the chair and sit down. Walk at his or her regular pace. Start timing on the word "go" and stop timing when the subject is seated again correctly in the chair with their back resting on the back of the chair. Interpretation: <10 seconds is normal, <20 seconds is good mobility, can go out alone, mobile without a gait aid and <30 seconds = problems, cannot go outside alone, requires a gait aid.
Sit to stand | From enrollment to the end of treatment at 10 weeks
  It counts the number of times the patient comes to a full standing position in 30 seconds. Record the number of times the patient stands in 30 seconds. An average score indicates a risk for falls: adjusted by age group and gender the scores ranges from less than 14 or less than 4.
6-minute walk test | From enrollment to the end of treatment at 10 weeks
  The 6-minute walk test (6MWT) is an assessment to determine a person's exercise tolerance. It is a low risk test that measures how far a person can walk in 6 minutes. It may be useful for measuring the functional ability and fitness of people with certain health conditions. Evidence suggests that the minimum score for healthy adults is 400 m. Scoring less than 400 meters suggests reduced exercise capacity.

CONTACTS AND LOCATIONS:
Overall Officials: Pere Roura-Poch, PhD, Principal Investigator — Vic Hospital Consortium
Locations (1):
- Health and Welfare Sciences School, Vic, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
The principal investigator will provide participant data if a justified request is received.
Supporting Information: CSR
Time Frame: 5 years after completion
Access Criteria: Adressing a letter with objectives and a justification about data needed